CLINICAL TRIAL: NCT00052923
Title: Randomized Phase III Trial Of Rituximab (NSC #687451) And Autologous Stem Cell Transplantation For B Cell Diffuse Large Cell Lymphoma
Brief Title: Stem Cell Transplantation With or Without Rituximab in Treating Patients With Relapsed or Progressive B-Cell Diffuse Large Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000258802; ECOG-E2499; CALGB-50205; CALGB-E2499
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-06

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Filgrastim; Rituximab; Carmustine; Cyclophosphamide; Etoposide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: carmustine
Drug: cyclophosphamide
Drug: etoposide
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Monoclonal antibodies, such as rituximab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether stem cell transplantation is more effective with or without rituximab in treating relapsed or progressive B-cell diffuse large cell lymphoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of stem cell transplantation with or without rituximab in treating patients who have relapsed or progressive B-cell diffuse large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival of patients with relapsed or progressive B-cell diffuse large cell lymphoma undergoing stem cell transplantation with or without post-transplant rituximab.
* Evaluate the effect of rituximab, administered post-transplant, on the procedure-related mortality of these patients.
* Determine the potential infectious complications of the addition of this drug to autologous stem cell transplantation in these patients.
* Compare overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to relapse (relapsed more than 6 months after either initial complete remission [CR] or CR with positive positron emission tomography or MRI [gallium] vs failed to achieve initial CR or relapsed within 6 months after either initial CR or CR with positive PET or MRI [gallium]) and prior rituximab (yes vs no).

Stem cell mobilization

* Patients receive rituximab IV over 4-8 hours on days 1 and 5. Patients also receive cyclophosphamide IV over 2 hours on day 8 and filgrastim (G-CSF) subcutaneously (SC) beginning on day 9 and continuing until the last day of apheresis. Stem cells are collected over 1-3 days.

Preparative regimen

* Regimen A (patients who have received prior radiotherapy or are ≥ 61 years of age): Patients receive carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 2 hours on day -2.
* Regimen B (all other patients): Patients undergo total body irradiation twice daily on days -8 to -5. Patients receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 2 hours on day -2.

Stem cells are reinfused on day 0. Patients are then randomized to one of two post-transplant treatment arms.

Post-transplant treatment

* Arm I (rituximab): Patients receive G-CSF SC beginning on day 6 and continuing until blood counts recover. Patients receive rituximab IV over 4-8 hours every 7 days for 4 doses, starting on day 45 post-transplant. Course of rituximab is repeated beginning on day 180 post-transplant.
* Arm II (no rituximab): Patients receive G-CSF as in arm I. Patients are followed for 10 years.

PROJECTED ACCRUAL: A total of 427 patients will be accrued for this study within 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large cell lymphoma and meeting the following criteria:

  * B-cell type with expression of CD20 either at diagnosis or at relapse
  * Relapse after having achieved an initial complete remission (CR) or failure to achieve initial CR (residual radiographic abnormalities after primary therapy allowed if these abnormalities are also positive by positron emission tomography or MRI [gallium])
  * No newly diagnosed disease
* No progressive or stable disease to most recent salvage therapy

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST or ALT < 3 times upper limit of normal

Renal

* Creatinine ≤ 2.0 mg/dL OR
* Creatinine clearance ≥ 40 mL/min

Cardiovascular

* Cardiac ejection fraction ≥ 40%

Pulmonary

* DLCO ≥ 60% of predicted

Other

* No other malignancy within the past 2 years except basal cell skin cancer or carcinoma in situ of the cervix
* No active infection requiring oral or IV antibiotics
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* No more than 3 prior immunotherapy regimens

Chemotherapy

* No more than 3 prior chemotherapy regimens

  * Addition of radiation or a monoclonal antibody to chemotherapy is considered one treatment regimen if the addition was part of the initial treatment plan
  * Addition of these therapies due to lack of response or poor response would be considered an additional treatment regimen whether given in front-line or salvage setting

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* No more than 3 prior radiotherapy regimens
* No prior radioimmunotherapy

Surgery

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2003-03; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Procedure-related mortality
Overall survival
Potential infectious complications of the addition of rituximab to autologous stem cell transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Charles A. Linker, MD, Study Chair — University of California, San Francisco